CLINICAL TRIAL: NCT00176202
Title: Controlled Trial of Risperidone and Divalproex Sodium With MRI Assessment of Affected Circuitry in Pre and Post Treatment in Pediatric Bipolar
Brief Title: Risperidone and Divalproex Sodium With MRI Assessment in Pediatric Bipolar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mani Pavuluri, Director of BRAIN Center, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIS-BIP-407
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Anticonvulsants; Risperidone; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone (Active Comparator): Risperidone is an antimanic medication and is a second generation antipsychotic
  Interventions: Drug: risperidone
- Divalproex sodium (Active Comparator): Divalproex sodium is an antiepileptic medication and is a mood stabilizer
  Interventions: Drug: Divalproex Sodium

INTERVENTIONS:
Drug: Divalproex Sodium — Divalproex sodium is a mood stabilizer
  Other Names: antiepileptic; valproic acid
  Arms: Divalproex sodium
Drug: risperidone — Risperidone is a second generation antipsychotic and antimanic drug
  Other Names: antipsychotic; risperdal
  Arms: Risperidone

SUMMARY:
The study is to examine the null hypothesis that risperidone and divalproex sodium are equally effective in treating/stabilizing pediatric bipolar disorder.

DETAILED DESCRIPTION:
Pediatric Bipolar Disorder (PBD) severely impairs a child's emotional development, and is associated with alarming rates of suicide, school failure, aggression, risk taking behaviors and substance abuse (Geller et al, 1998; 2001; Carlson et al, 1998). At present, very little is known about the pathophysiology or optimal treatment of PBD. The long range goals of this proposal are threefold: to investigate a range of pharmacotherapeutic agents that are safe and efficacious for PBD, to use fMRI techniques to examine abnormalities in brain function in this disorder, as well as any change in brain function after treatment.

In contrast to the adult literature, we are aware of only two prospective studies assessing the efficacy of standard mood stabilizers in a pediatric sample. In one, lithium was found to be moderately effective in PBD with comorbid substance abuse (Geller et al, 1998). In the other, divalproex sodium, lithium and carbamazepine produced a maximum of 50% symptom reduction (Kowatch et al, 2000). Subsequently, Kafantaris et al (2001) observed a potentiation of lithium's antimanic effect when combined with risperidone. Further, a prospective, open trial of olanzapine for PBD reported a 70% symptom reduction (Frazier et al, 2001) with a retention rate of 96% compared to only 7% with classic mood stabilizers (Kowatch et al, 2000).

Thus, parallelling adult studies (Sachs et al, 2000), novel antipsychotics are a promising treatment in this population. Further, up to 60% of acute PBD episodes present with psychotic features (Geller et al, in press). Finally, the time to full effect with mood stabilizers is often 4 weeks in children (Kowatch et al, 2000; Geller et al, 1998; Kafantaris et al, 2001), whereas antipsychotics usually have a more rapid response onset (Pavuluri et al, in press). Given the potential efficacy of novel antipsychotics for PBD, the aim is to conduct a randomized trial comparing a novel antipsychotic to a standard mood stabilizer:

ELIGIBILITY:
Inclusion Criteria:

* Children with Bipolar Disorder
* Must be able to swallow tablets

Exclusion Criteria:

* Children with general medical condition such as head injury, epilepsy, endocrine disorders
* Those who are on mood altering medications such as steroids, and those diagnosed with mental retardation are excluded to avoid confounding and contributing factors to mood swings.
* If we discover during the interview that the parent and/or child does not understand the consent/assent procedures, we will exclude them.

We expect only a small number of children to be excluded from the study due to exclusionary criteria. Selection of the subjects is not based on sex, race, or ethnic group.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2003-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mani Pavuluri, MD, Principal Investigator — University of Ilinois at Chicago
Locations (3):
- United States (3):
  - Neuro Psychiatric Institute (NPI), Chicago, Illinois
  - NPI, University of Illinois at Chicago, Chicago, Illinois
  - NPI, Chicago, Illinois

REFERENCES:
- [Derived] Pavuluri MN, Passarotti AM, Fitzgerald JM, Wegbreit E, Sweeney JA. Risperidone and divalproex differentially engage the fronto-striato-temporal circuitry in pediatric mania: a pharmacological functional magnetic resonance imaging study. J Am Acad Child Adolesc Psychiatry. 2012 Feb;51(2):157-170.e5. doi: 10.1016/j.jaac.2011.10.019. Epub 2011 Dec 23. PMID 22265362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment :From Sep2005 - Jan 2008.in Clinic Subjects enrolled:65
Pre-assignment Details: Exclusion Criteria:
  * Children with general medical condition such as head injury, epilepsy, endocrine disorders
  * Those who are on mood altering medications such as steroids, and those diagnosed with mental retardation are excluded to avoid confounding and contributing factors to mood swings.
Groups:
- Risperidone: The study aimed to compare the antipsychotic medication i.e., risperidone's efficacy with that of divalproex sodium (which is an antiepileptic medication) in treating/stabilizing pediatric bipolar disorder.
- Divalproex Sodium: This is antiepileptic medication and is a comparator drug to see if it is as efficacious as risperidone assumption is both have equal efficacy with no difference between the two.
Period: Overall Study
Arm/Group | Risperidone | Divalproex Sodium
Started | 32 | 33
Completed | 27 | 17
Not Completed | 5 | 16

BASELINE CHARACTERISTICS:
Population: AGE 10 TO 20 YRS GENDER :BOTH
Groups:
- Risperidone: Risperidone is an antipsychotic medication and is used to treat mania. Its trade name is Risperdal.
  Aim of the study is to cross compare the relative efficacy and safety of risperidone and divalproex sodium in treating/stabilizing mania in pediatric bipolar disorder.
- Divalproex: Divalproex sodium, also referred to as divalproex is an antiepileptic medication used for mania and is referred to as mood stabilizer. Its trade name is Depakote.
- Total: Total of all reporting groups
Arm/Group | Risperidone | Divalproex | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.47 (3.18) | 11.23 (3.50) | 10.85 (3.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: This measure has 11 items. The purpose of each item is to rate the severity of that abnormality in the patient. A severity rating is assigned to each of the eleven items, based on the patient's subjective report of his or her condition over the previous forty-eight hours and the clinician's behavioral observations during the interview, with the emphasis on the latter. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Total score of zero to 60 is possible, zero being normal and 60 being severe, 12 serving as a cut off point for illness if equal or above. There are several ways to show change in outcome. We show the mean and standard deviation at week 0 and 6.
Time Frame: Six week study with assessment at baseline and end of the study (at the end of 6 weeks or earlier if they ended the study before 6 week end point).
Population: Inclusion criteria were a DSM-IV diagnosis of bipolar disorder Type I (mixed or manic episode); 8 to 18 years old; and medication free or currently clinically unstable on medication, justifying termination of the ineffective regimen.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Divalproex: Divalproex was titrated up to 15 mg/kg/day over 3 days and serum level was measured at the end of 5 days. Divalproex dose was immediately adjusted on obtaining the serum level to aim for 80-120 μg/ml- trough, while ensuring that the dose was tolerated when increased. Serum valproate level was repeated at the end of the study.
- Risperidone: Risperidone was initiated at 0.25 mg to 0.50 mg per day. The dose was titrated to a maximum of 2 mg per day by increments of 0.25-0.5 mg every 2 days to achieve a maximum tolerable level by day 7.
Arm/Group | Divalproex | Risperidone
Number analyzed (Participants) | 33 | 32
units on a scale
  Baseline | 25.09 (7.51) | 30.59 (7.04)
  Last observation carried forward (LOCF) | 15.24 (12.49) | 10.22 (10.50)
Statistical Analysis 1: Comparison: Divalproex; Test type: Superiority or Other; p < 0.01, Chi-squared
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p < 0.01, Chi-squared

2. Secondary Outcome: Child Depression Rating Scale- Revised (CDRS-R)
Description: Response for depressive symptoms was defined as a score less than 40 on the CDRS-R. Range is 18 to 120. Score 18 is normal and higher score signifies depression. The Children's Depression Rating Scale (CDRS) is a 16-item measure used to determine the severity of depression in children 6-18 years of age. Items are measured on 3-, 4-, 5-, and 6-point scales. The mean and standard deviation are measured in this study to illustrate outcome at baseline and when the subject ended the study.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex | Risperidone
Number analyzed (Participants) | 33 | 32
units on a scale
  Baseline | 40.76 (13.34) | 41.72 (17.44)
  Last Observation Carried Forward (p<.01) | 35.76 (15.01) | 25.88 (9.13)
Statistical Analysis 1: Comparison: Divalproex; Test type: Superiority or Other; p < .01, Chi-squared
Statistical Analysis 2: Comparison: Risperidone; Test type: Superiority or Other; p = 0.01, Chi-squared

3. Secondary Outcome: Child Mania Rating Scale (CMRS)
Description: Child Mania rating scale is a parent rated measure to screen for symptoms of mania. It includes 21 items reflecting the DSM-IV criteria for a manic episode. Each item is answered on a four-point Likert type scale anchored by 0 (Never/Rare), 1 (Sometimes), 2 (Often), and 3 (Very Often). Maximum score possible is 63. Score higher than 20 is considered clinically significant, and this is a dimensional score of manic severity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- Risperidone: Antipsychotic medication used as a anti manic agent
- Divalproex Sodium: Antiepileptic medication used as mood stabilizer/antimanic agent
Arm/Group | Risperidone | Divalproex Sodium
Number analyzed (Participants) | 32 | 33
units on scale
  Baseline | 30.84 (10.87) | 28.0 (9.02)
  LOCF | 16.35 (13.09) | 19.20 (12.66)
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority or Other; p < 0.01, Chi-squared — In case of both risperidone and divalproex sodium; effect size = -1.59
Statistical Analysis 2: Comparison: Divalproex Sodium; Test type: Superiority or Other; p < 0.01, Chi-squared; Effect size = -1.33

4. Secondary Outcome: Clinical Global Improvement in Bipolar Disorder Overall (CGI-BP Overall)
Description: Severity of Illness and Global Improvement are rated on a 7-point scale by the clinician. In addition to rating the overall illness with the CGI-BP, severity and improvement are considered on various other dimensions such as mania, depression, attention deficit/hyperactivity, psychosis, aggression and sleep difficulties. Score of 1, 2 and 3 would mean there is clinically observed symptom improvement where 1 is the best outcome than 2 or 3. The point 4 is the point where the subject presents at baseline of that specific individual. If they become worse on clinical symptoms, they are rated as 5, 6 or 7 where 7 is worse than 5.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Divalproex Sodium
Number analyzed (Participants) | 32 | 33
units on a scale
  Baseline | 4.80 (1.06) | 4.37 (0.67)
  LOCF | 2.77 (1.28) | 2.97 (1.50)
Statistical Analysis 1: Comparison: Risperidone; baseline is compared to LOCF to determine the p value; Test type: Superiority or Other; p < 0.01, Chi-squared
Statistical Analysis 2: Comparison: Divalproex Sodium; Test type: Superiority or Other; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: Weekly from baseline and for 6 weeks; 7 waves of data.
Groups:
- Risperidone: Likely side effects include weight gain, muscle stiffness, sedation and tiredness.
  Clarification: We did not note any serious side effects with either drug. We reported any adverse event that is found in greater than 5% of the participants in each group. Frequency of adverse events do not equal the fact that they are serious adverse events at any individual level.
- Depakote or Divalproex Sodium: Likely side effects include gastrointestinal side effects such as stomach discomfort, weight gain, agitation and sedation, fatigue or tiredness.
  Clarification: We did not note any serious side effects with either drug. We reported any adverse event that is found in greater than 5% of the participants in each group. Frequency of adverse events do not equal the fact that they are serious adverse events at any individual level.
Arm/Group | Risperidone | Depakote or Divalproex Sodium
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 8/32 | 10/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=32) | Depakote or Divalproex Sodium (N=33)
Increased appetite (Metabolism and nutrition disorders) | 8 (8) | 10 (10)
Irritable/agitated (Nervous system disorders) | 0 (0) | 7 (7)
stomach discomfort (Gastrointestinal disorders) | 6 (6) | 5 (5)
sleepiness (Nervous system disorders) | 5 (5) | 4 (4)
fatigue/tiredness (Nervous system disorders) | 5 (5) | 4 (4)
insomnia (Nervous system disorders) | 0 (0) | 4 (4)
weight gain (Metabolism and nutrition disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes